CLINICAL TRIAL: NCT04643639
Title: An Open-label Randomized Controlled Experimental Endotoxemia Study on the Effects of the Cytokine-adsorber CytoSorb on the Development of Immunoparalysis in Humans
Brief Title: Assessing the Effects of CytoSorb Hemoperfusion on the Development on Immunoparalysis
Acronym: EndoSorb
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The EndoSorb Study
Record Dates: First submitted 2020-09-15; First posted 2020-11-25 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2021-03

CONDITIONS: Sepsis; Immune Deficiency; Hemoperfusion; Blood Purification
MeSH Terms: conditions — Sepsis; Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Device: CytoSorb hemoperfusion
- Control (No Intervention)

INTERVENTIONS:
Device: CytoSorb hemoperfusion — Subjects will be treated with CytoSorb hemoperfusion (in stand-alone setup) for 6 hours at a flow rate of 250 ml/min during endotoxemia.
  Arms: Active

SUMMARY:
In this randomized, open-label study, the investigators will assess whether CytoSorb hemoperfusion will prevent or attenuate the development of immunoparalysis in healthy volunteers undergoing repeated experimental endotoxemia.

DETAILED DESCRIPTION:
Sepsis is an inflammatory syndrome with high mortality rates and increasing incidence. Sepsis-induced immunoparalysis, increasingly recognized as the overriding immune disorder in sepsis patients, attributes significantly to late mortality in sepsis patients.

The investigators hypothesize that 'blood purification' techniques targeted at the removal of excess circulating cytokines, such as the CytoSorb hemoperfusion device, might prevent or attenuate the development of immunoparalysis.

The objective of this trial is to determine the effects of CytoSorb hemoperfusion on the development of immunoparalysis in a repeated experimental endotoxemia model in healthy male volunteers.

To this end, 24 healthy male volunteers subjects will be randomized in a 1:1 fashion into one of two treatment groups (active or control). Both study groups will undergo two endotoxin challenges, separated by seven days. To this end, endotoxin (LPS) will be administered as a bolus of 1 ng/kg, followed by continuous infusion of 0.5 ng/kg/hr for three hours. The active group will be treated with CytoSorb hemoperfusion during the first endotoxin challenge, whereas the control group will receive no additional treatment. During both endotoxin challenges, blood samples will be obtained serially to measure levels of circulating cytokines and other inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Male
* Age ≥ 18 and ≤ 35 years
* Healthy (as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) and routine clinical laboratory parameters)

Exclusion Criteria:

* Use of any medication
* Smoking
* Known anaphylaxis or hypersensitivity to any (non-)investigational products or their excipients.
* History or signs of atopic syndrome (asthma, rhinitis with medication and/or eczema)
* History or signs of hematological disease
* History or signs of thromboembolic disorders
* History of (intracranial) aneurysmal or hemorrhagic diseases
* History of heparin-induced thrombocytopenia (HIT)
* Thrombocytopenia (<150*109/ml) or anemia (hemoglobin < 8.0 mmol/L)
* History, signs or symptoms of cardiovascular disease, in particular:

  * Previous spontaneous vagal collapse
  * History of atrial or ventricular arrhythmia
  * Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrio-ventricular block or a complete left bundle branch block
  * Hypertension (defined as RR systolic > 160 or RR diastolic > 90 mmHg)
  * Hypotension (defined as RR systolic < 100 or RR diastolic < 50 mmHg)
* Renal impairment (defined as plasma creatinine >120 μmol/l)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Medical history of any disease associated with immune deficiency
* Signs of infection (CRP > 20 mg/L, WBC > 12x109/L or < 4x109/L)
* Clinically significant acute illness, including infections or trauma, within 1 month of the first endotoxin challenge
* Previous (participation in a study with) endotoxin (LPS) administration
* Any vaccination within 3 months within of the first endotoxin challenge
* Participation in a drug trial or donation of blood within 3 months prior to first endotoxin challenge
* Recent hospital admission or surgery with general anesthesia within 3 months prior to first endotoxin challenge
* Use of recreational drugs within 1 month of the first endotoxin challenge
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Between group differences in plasma interleukin (IL)-6 levels during the second endotoxin challenge. | Samples will be obtained starting 1 hour prior until 8 hours after endotoxin administration
  Blood samples will be obtained at predefined time points before, during and after endotoxin administration to assess plasma levels (in pg/mL) of circulating inflammatory mediatiors. To assess between group differences, the area under the curve (AUC) of the time concentration curve (expressed in arbitrary units) of each inflammatory mediator will be calculated.

SECONDARY OUTCOMES:
Between group differences in plasma levels of other inflammatory cytokines during the second endotoxin challenge. | Samples will be obtained starting 1 hour prior until 8 hours after endotoxin administration
  Interleukin (IL)-6, IL-8, IL-10, Monocyte Chemoattractant Protein (MCP)-1, C-X-C motif chemokine ligand (CXCL)-10, Macrophage Inflammatory Protein (MIP)-1α, MIP-1β, and Granulocyte Colony-Stimulating Factor (G-CSF)
Between group differences in mHLA-DR expression | 1 hour before, 3 hours after and 6 hours after endotoxin administration
  Differences in Human Leukocyte Antigen (HLA)-DR expression on monocytes will be assessed using flowcytometry.
Between group differences in norepinephrine sensitivity | One hour before and 4 hours after endotoxin administration during the first endotoxin challenge
  To assess the effects of CytoSorb hemoperfusion on norepinephrine sensitivity, norepinephrine will be administered in increasing dosages (0.025; 0.05 and 0.1 γ) for 5 minutes per dose. Blood pressure will be recorded continuously with an arterial catheter.
Cytokine clearance by the adsorber | Every 30 minutes until cessation of hemoperfusion (six hours after endotoxin administration)
  Blood samples will be obtained from the afferent and efferent tubing of the CytoSorb adsorber to calculate clearance of cytokines by the adsorber
Between group differences in endotoxemia-induced metabolic activity of platelets | 1 hour prior until 8 hours after endotoxin administration
  Blood samples will be collected in citrated tubes to allow assessment of ATP production by platelets.
Between group differences in endotoxemia-induced clinical symptoms | Every 30 minutes from 1 hour prior until 8 hours after endotoxin administration
  Clinical symptoms will be scored on a Likert scale (ranging from 0 to 5) in a composite endpoint consisting of headache, nausea, shivering, muscle soreness and lower back pain. Higher numbers indicate more severe symptoms.
Between group differences in body temperature | Every 30 minutes from 1 hour prior until 8 hours after endotoxin administration
  Body temperature will be assessed using tympanic temperature measurements
Between group differences in blood pressure | From 1 hour prior until 8 hours after endotoxin administration
  Systolic, diastolic and mean arterial pressure will be measured continuously using a radial artery catheter.
Between group differences in heart rate | From 1 hour prior until 8 hours after endotoxin administration
  Heart rate will be recorded continuously using a 3-lead ECG.
Between group differences in markers of endothelial injury | Samples will be obtained starting 1 hour prior until 8 hours after endotoxin administration
  Vascular cell adhesion protein (VCAM)-1 and Intercellular Adhesion Molecule (ICAM)-1

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jansen A, Waalders NJB, van Lier DPT, Kox M, Pickkers P. CytoSorb hemoperfusion markedly attenuates circulating cytokine concentrations during systemic inflammation in humans in vivo. Crit Care. 2023 Mar 21;27(1):117. doi: 10.1186/s13054-023-04391-z. PMID 36945034